CLINICAL TRIAL: NCT02587884
Title: Anti-recurrence Treatment of Postresection on Hepatocellular Carcinoma Patients With Microvascular Invasion Presence and Over-expression of Aspartate Beta-hydroxylase: A Randomized Controlled Study
Brief Title: Anti-recurrence Treatment of Postresection on HCC Patients With MVI Presence and Over-expression of ASPH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital Affiliation: Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2015-01-024
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Recurrence; Microvascular Invasion; Aspartate beta-hydroxylase
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group TACE (Active Comparator): Patients will treated with TACE after resection.
  Interventions: Procedure: TACE
- Group Control (No Intervention): Patients will treated without TACE after resection.

INTERVENTIONS:
Procedure: TACE — Patients will treated by TACE in 4 or 8 weeks after operation.
  Other Names: Transhepatic Arterial Chemotherapy And Embolization
  Arms: Group TACE

SUMMARY:
The aim of this study is to explore the effect of Transarterial Chemoembolization (TACE) on the prognosis of patients with microvascular invasion presence(MVI) and overexpression of Aspartate-β-hydroxylase(ASPH).

ELIGIBILITY:
Inclusion Criteria:

1. Via clinical diagnosis and confirm it is primary liver cancer
2. Pathological evidence of HCC
3. Confirm presence of MVI and over-expression of ASPH after opreation
4. Within Milan criteria
5. Estimate tumor can gain treatment of curing operation
6. No evidence for extrahepatic metestasis
7. liver function ：Child-Pugh A/B

Exclusion Criteria:

1. Reject to attend
2. Impossible to come to our hospital for physical examination regularly
3. Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction
4. Female with pregnancy or during the lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Time to recurrence | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China